CLINICAL TRIAL: NCT06160323
Title: Upfront Endoscopic Ultrasound-guided Celiac Ganglion Neurolysis Versus Conventional Step-up Approach for Patients With Painful, Inoperable Pancreatic Cancer
Brief Title: Upfront EUS CGN/CPN vs Conventional Step up Approach for Inoperable Painful Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023.294
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer Non-resectable; Tumor Pancreas; Pain Cancer
Keywords: Pancreatic Cancer Non-resectable; tumor pain; endoscopic ultrasound-guided celiac ganglion neurolysis
MeSH Terms: conditions — Pancreatic Neoplasms; Cancer Pain

STUDY DESIGN:
Intervention Model Description: Patient will be randomly assigned in a 1:1 ratio to either the upfront EUS-guided CGN/CPN approach or to the conventional step-up approach at the time of EUS. Site-specific block randomization will be performed via an online web-based randomization program with a concealed, fixed block size.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will be masked on their randomization until (i) 3 month from randomization (study endpoint) or (ii) after 4 weeks if VAS score >= 7 or VAS score fails to improve by 20% despite optimal oral analgesics, when they will be allowed to opt for EUS-guided CGN/ CPN. The pain assessment will be performed by assessors who are blinded to the randomized group each time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided coeliac ganglion neurolysis / celiac plexus neurolysis (Active Comparator): Patient would undergo a EUS diagnostic procedure with or without a biopsy. Patient would be blinded to the group they were assigned. The procedure will be performed with a linear array echoendoscope (EUS) under conscious sedation or monitored anaesthesia care.
  For cases in which celiac ganglia could not be visualized, EUS-guided coeliac plexus neurolysis (CPN) will be performed.
  Interventions: Procedure: EUS-guided coeliac ganglion neurolysis / celiac plexus neurolysis
- Conventional step-up approach (Active Comparator): Patient would undergo a EUS diagnostic procedure with or without a biopsy. Patient would be blinded to the group they were assigned. The concept of the conventional step-up approach is to follow ESMO clinical practice guidelines for cancer pain.
  In case of inadequate pain control, the analgesics will be stepped up according to the guidelines. After 4 weeks, if patient's VAS score more than 7 or VAS score fails to improve by 20% despite optimal oral analgesics, patients are given the option of EUS-guided CGN/ CPN.
  Interventions: Procedure: EUS-guided coeliac ganglion neurolysis / celiac plexus neurolysis

INTERVENTIONS:
Procedure: EUS-guided coeliac ganglion neurolysis / celiac plexus neurolysis — The EUS scope was first inserted into the stomach, and the coeliac trunk was visualized by scanning from the lesser curve of the gastric body. After visualization, the scope was rotated clockwise, enabling visualization and identification of the left adrenal gland. The coeliac ganglia are often seen to the left of the coeliac artery, between the aorta and the left adrenal gland, at the level between the coeliac artery and the left adrenal artery. They are also visualized cephalad to the coeliac artery in some cases. Hypoechoic nodular structures linked by hypoechoic threads residing in the periphery of this region were defined as the coeliac ganglia . A 19G or 22G needle was used for puncture of the CGN. After confirming the lack of backflow of blood with aspiration, a mixture of 5ml of 0.25-0.5% bupivacaine and 5ml absolute alcohol was injected.
  For cases in which celiac ganglia could not be visualized, EUS-guided coeliac plexus neurolysis (CPN) will be performed.

SUMMARY:
Patients with unresectable pancreatic cancer are often demoralized by intractable, persistent and incapacitating pain. It must be managed aggressively and strong opioids are recommended as the mainstay of treatment. However, patients develop opioid-related adverse effects. EUS-guided celiac plexus neurolysis (CPN) and celiac ganglion neurolysis (CGN) has been shown to provide high efficacy for pain control. The optimal timing, however, is in debate.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years old
2. Diagnosed to have inoperable pancreatic cancer
3. Presence of tumor pain (centrally located, constant, with no other obvious cause) with a VAS >= 3
4. Karnofsky performance status >= 60
5. Planned for EUS examination and/or biopsy of the pancreatic tumor

Exclusion Criteria:

1. Allergy to bupivacaine, or alcohol
2. Potentially operable after neoadjuvant therapy
3. Expected survival of less than 3 months
4. Patient who is already on opioids for pain control
5. Previous percutaneous or EUS-guided CGN/ CPN
6. Recurrent pancreatic tumors after operation
7. Uncorrectable coagulopathy
8. Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The mean change in VAS pain score at 3 months | 3 months
  The mean change in VAS pain score at 3 months when compared to baseline (pre-procedure) between upfront EUS group and conventional step-up group

SECONDARY OUTCOMES:
The mean percentage and absolute change in VAS pain score at 1 month | 1 month
  The mean percentage and absolute change in VAS pain score at 1 month when compared to baseline (pre-procedure)
The mean percentage in VAS pain score at 3 month | 3 months
  The mean percentage in VAS pain score at 3 month when compared to baseline (pre-procedure)
Short form McGill Pain Questionnaire-2 | 3 months
  The absolute and mean percentage change in Short form McGill Pain Questionnaire-2
Brief Pain Inventory | 3 months
  The absolute and mean percentage change in Brief Pain Inventory
Morphine equivalent (MEQ) consumption | 3 months
  Absolute use and percentage change of morphine (expressed in morphine equivalent (MEQ) consumption) when compared to baseline
Common opioid-related adverse effects | 3 months
  Common opioid-related adverse effects including nausea, pruritus, constipation and drowsiness will be recorded
Quality of life | 3 months
  Changes of the score in quality of life (EORTC QLQ-C30)
Karnofsky performance status | 12 weeks
  Karnofsky performance status at baseline, 4 weeks, 8 weeks and 12 weeks
Adverse events from the EUS-guided CGN/CPN | 7 days
  Adverse events from the EUS-guided CGN/CPN will be recorded
Breakthrough visits | 4 weeks
  Breakthrough visits in between the 4 weeks
Need for and timing EUS-guided CGN/CPN for the conventional group | 3months
  Need for and timing EUS-guided CGN/CPN for the conventional group will be recorded
Overall survival | 48 weeks
  Date of death will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong